CLINICAL TRIAL: NCT04210947
Title: Effects of Different Variation of Myofascial Release Application Speed on Muscle Mechanical Properties
Brief Title: Effect of Foam Rolling on Muscle Mechanical Properties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Atilla Çağatay Sezik, PhD. Student, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Sporcufoamroller
Record Dates: First submitted 2019-12-22; First posted 2019-12-26 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Sports Physical Therapy
Keywords: sports physiotherapy; self-myofascial release; foam-roller; muscle biomechanical properties

STUDY DESIGN:
Intervention Model Description: Participants will use a foam roller at three different paces in a randomized sequence with a week between,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Foam-roller I-II-III (Experimental): Participants will use foam roller in following order of 30RPM(I), 15RPM(II) and self-determined(III)
  Interventions: Other: 30 rolls per minute(30RPM); Other: 15 rolls per minute(15RPM); Other: self-determined
- Foam-roller I-III-II (Experimental): Participants will use foam roller in following order of 30RPM(I), self-determined(III) and 15RPM(II)
  Interventions: Other: 30 rolls per minute(30RPM); Other: 15 rolls per minute(15RPM); Other: self-determined
- Foam-roller II-I-III (Experimental): Participants will use foam roller in following order of 15RPM(II), 30RPM(I) and self-determined(III)
  Interventions: Other: 30 rolls per minute(30RPM); Other: 15 rolls per minute(15RPM); Other: self-determined
- Foam-roller II-III-I (Experimental): Participants will use foam roller in following order of 15RPM(II), self-determined(III) and 30RPM(I)
  Interventions: Other: 30 rolls per minute(30RPM); Other: 15 rolls per minute(15RPM); Other: self-determined
- Foam-roller III-I-II (Experimental): Participants will use foam roller in following order of self-determined(III), 30RPM(I) and 15RPM(II)
  Interventions: Other: 30 rolls per minute(30RPM); Other: 15 rolls per minute(15RPM); Other: self-determined
- Foam-roller III-II-I (Experimental): Participants will use foam roller in following order of self-determined(III), 15RPM(II) and 30RPM(I)
  Interventions: Other: 30 rolls per minute(30RPM); Other: 15 rolls per minute(15RPM); Other: self-determined

INTERVENTIONS:
Other: 30 rolls per minute(30RPM) — Participants will start using foam roller from muscle origin to insertion with a speed of 2 secs. Then comeback from insertion to origin with 2 secs. With total of 15 repeats x 2 sets per leg. With 30 seconds rest between.
Other: 15 rolls per minute(15RPM) — Participants will start using foam roller from muscle origin to insertion with a speed of 4 secs. Then comeback from insertion to origin with 4 secs. With total of 15 repeats x 2 sets per leg. With 30 seconds rest between.
Other: self-determined — Participants will start using foam roller from muscle origin to insertion with self determined-speed. Then comeback from insertion to origin with same pace. With total of 15 repeats x 2 sets per leg. With 30 seconds rest between.

SUMMARY:
This study evaluates effect of self-myofascial release in different paces on muscle biomechanics. All participants will use foam roller in different paces once in a week with weeks apart.

DETAILED DESCRIPTION:
Foam-roller is a widely used self-myofascial release method in sports. Although, effects of foam-roller has been shown, there is no defined speed of usage. Using foam-roller in different paces could cause different changes.

ELIGIBILITY:
Inclusion Criteria:

* Being a professional athlete with at least 2 years of sport history

Exclusion Criteria:

* Having a chronic-systemic disease
* Having a lower extremity injury

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2022-10-16 (Actual); Study Completion 2023-04-16 (Actual)

PRIMARY OUTCOMES:
Viscoelastic measurement Change | baseline and 15 minutes
  Myotonometer-3 will be used for measuring viscoelastic properties (tone, elasticity, stiffness)

SECONDARY OUTCOMES:
Hip Flexors Tightness | baseline and 15 minutes
  Modified Thomas test would be used for measuring hip flexors tightness

CONTACTS AND LOCATIONS:
Overall Officials: Atilla Çağatay Sezik, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Curran PF, Fiore RD, Crisco JJ. A comparison of the pressure exerted on soft tissue by 2 myofascial rollers. J Sport Rehabil. 2008 Nov;17(4):432-42. doi: 10.1123/jsr.17.4.432. PMID 19160916
- [Background] Kumka M, Bonar J. Fascia: a morphological description and classification system based on a literature review. J Can Chiropr Assoc. 2012 Sep;56(3):179-91. PMID 22997468
- [Background] Chaitow L. Somatic dysfunction and fascia's gliding-potential. J Bodyw Mov Ther. 2014 Jan;18(1):1-3. doi: 10.1016/j.jbmt.2013.11.019. Epub 2013 Dec 3. No abstract available. PMID 24411142
- [Background] Stecco A, Meneghini A, Stern R, Stecco C, Imamura M. Ultrasonography in myofascial neck pain: randomized clinical trial for diagnosis and follow-up. Surg Radiol Anat. 2014 Apr;36(3):243-53. doi: 10.1007/s00276-013-1185-2. Epub 2013 Aug 23. PMID 23975091
- [Background] Stecco C, Stern R, Porzionato A, Macchi V, Masiero S, Stecco A, De Caro R. Hyaluronan within fascia in the etiology of myofascial pain. Surg Radiol Anat. 2011 Dec;33(10):891-6. doi: 10.1007/s00276-011-0876-9. Epub 2011 Oct 2. PMID 21964857
- [Background] MacDonald GZ, Penney MD, Mullaley ME, Cuconato AL, Drake CD, Behm DG, Button DC. An acute bout of self-myofascial release increases range of motion without a subsequent decrease in muscle activation or force. J Strength Cond Res. 2013 Mar;27(3):812-21. doi: 10.1519/JSC.0b013e31825c2bc1. PMID 22580977
- [Derived] Sezik AC, Uysal O, Firat T, Duzgun I, Bayrakci Tunay V. The Effects of Foam Rolling at Different Speeds on Mechanical Properties of Quadriceps Femoris. J Sports Sci Med. 2024 Sep 1;23(1):684-689. doi: 10.52082/jssm.2024.684. eCollection 2024 Sep. PMID 39228783